CLINICAL TRIAL: NCT01475630
Title: Randomised Controlled Trial on Physical Therapy PT) for TMJ Closed Lock
Brief Title: Physical Therapy for Temporomandibular Joint (TMJ) Closed Lock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, prof.dr. Antoon De Laat, Head of Service Dentistry, KU Leuven
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ML2210
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Disc Displacement, Without Reduction
Keywords: temporomandibular joint; rehabilitation medicine; joint diseases; physical therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Joint Diseases | interventions — Physical Therapy Modalities; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Other): information, avoiding parafunctions
  Interventions: Procedure: control
- physical therapy (Experimental): mobilisation, exercises ,..
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: physical therapy — mobilisation of the jaw, exercises, boostering information on avoiding parafunctions
  Other Names: physiotherapy
  Arms: physical therapy
Procedure: control — relaxation
  Other Names: counseling; information
  Arms: control

SUMMARY:
The aim of the present study was to investigate the effect of Physical Therapy (PT) on pain and mandibular function in patients with anterior disc displacement without reduction (ADD-R) or "closed lock" of the TMJ and this in a randomized controlled trial design.

DETAILED DESCRIPTION:
The study evaluated the effect of extra, technical PT over the traditional information on the benign nature of the disease and the advice to refrain from overuse or misuse of the masticatory system as in parafunctions.

ELIGIBILITY:
Inclusion Criteria:

* All patients were recruited from the Oral Pain and Dysfunction Clinic and strictly satisfied the RDC-TMD criteria for .for disc displacement without reduction with (group IIb) or without (group IIc) limitation of mouth opening, based upon history and clinical examination. Additionally, pain experienced during the first examination had to be ≥ 35mm on a visual analog scale (VAS) of 100mm.

Exclusion Criteria:

* Patients were excluded if their medical history mentioned orofacial traumata (contusion or fracture), systemic disorders (e.g. rheumatoid arthritis, fibromyalgia), cervical disorders (operationalized as complaints, pain or referral patterns of pain provoked during movements of the cervical spine), neurologic disorders (e.g. trigeminal neuralgia, migraine or tension type headache), drug or alcohol abuse, use of antidepressant or hormonal medication. Participants did not receive therapy for symptoms of TMD within the last 2 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-06; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
pain intensity | 1 year
  using VAS scales

SECONDARY OUTCOMES:
mouth opening | 1 year
  interincisal dstance measured by a ruler upon active and passive mouth opening
pressure pain threshold | 1 year
  the pressure pain threshold was measured using an algometer at the masseter and temporalis muscles bilaterally
mandibular function impairment questionnaire | 1 year
  Using a validated questionnaire the impact of the pain and limitaiton on normal masticatory function is monitored

CONTACTS AND LOCATIONS:
Overall Officials: Antoon De Laat, DDS,PhD, Principal Investigator — Catholic University Leuven
Locations (1):
- univ hospital sint Rafael, KULeuven, Leuven, Belgium

REFERENCES:
- [Derived] Craane B, Dijkstra PU, Stappaerts K, De Laat A. Randomized controlled trial on physical therapy for TMJ closed lock. J Dent Res. 2012 Apr;91(4):364-9. doi: 10.1177/0022034512438275. Epub 2012 Feb 8. PMID 22318373